CLINICAL TRIAL: NCT00921375
Title: Efficacy and Safety of TULY in Prevention and Treatment of Malignancy-associated Hyperuricemia
Brief Title: Safety and Efficacy of TULY (Rasburicase) in Prevention and Treatment of Malignancy-associated Hyperuricemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virchow Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VB037/2007; VB037 (Other: Protocol Number)
Record Dates: First submitted 2009-05-23; First posted 2009-06-16 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tuly, uric acid lowering drug (Experimental): TULY (rasburicase) 0.20 mg/kg body weight intravenously for 4 days
  Interventions: Drug: TULY

INTERVENTIONS:
Drug: TULY — TULY (rasburicase) 0.20 mg/kg body weight intravenously for 4 days

SUMMARY:
This study is a prospective, open-label, multicentre study. Hundred eligible patients with stage III or IV non-Hodgkin lymphoma (NHL) or acute lymphoblastic leukemia (ALL) with a peripheral white blood cell (WBC) count of > 25,000/µL or any leukemia or lymphoma with plasma uric acid level of at least 8 mg/dL will be treated with rasburicase 0.20 mg/kg body weight intravenously for 4 days. The primary endpoints viz., the percentage of reduction in plasma uric acid at 4 hrs after uric acid-lowering therapy, plasma uric acid AUC 0-96 hr and incidence of adverse events will be assessed during 11 days study period.

DETAILED DESCRIPTION:
All eligible patients will be treated with rasburicase 0.20 mg/kg body weight intravenously for 4 days. The primary endpoints viz., the percentage of reduction in plasma uric acid at 4 hrs after uric acid-lowering therapy, plasma uric acid AUC 0-96 hr and incidence of adverse events will be assessed during 11 days study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders aged between 1 to 75 years;
2. Patients with stage III or IV non-Hodgkin lymphoma (NHL) or acute lymphoblastic leukemia (ALL) with a peripheral WBC count of >25,000/µL or any leukemia or lymphoma with plasma uric acid level of at least 8 mg/dL;
3. Eastern Cooperative Oncology Group (ECOG) performance scale of ≤3;
4. Patients scheduled to receive chemotherapy.

Exclusion Criteria:

1. Patients with allergy or asthma, or hypersensitivity to urate oxidase, or hemolytic reactions;
2. Pregnant and lactating;
3. Patients with glucose-6-phosphate dehydrogenase deficiency;
4. Exposure to rasburicase or allopurinol within 7 days;
5. History of psychiatric or co-morbid unstable medical conditions

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage of reduction in plasma uric acid at 4 hrs after uric acid-lowering therapy | At the end of 4 hrs after initiation of uric acid lowering therapy; during 96 hrs of uric acid lowering therapy; Adverse events during the entire study period

SECONDARY OUTCOMES:
Plasma uric acid AUC 0-96 hr | At the end of 4 hrs after initiation of uric acid lowering therapy; during 96 hrs of uric acid lowering therapy; Adverse events during the entire study period
Incidence of adverse events | At the end of 4 hrs after initiation of uric acid lowering therapy; during 96 hrs of uric acid lowering therapy; Adverse events during the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Raghunadharao D, Principal Investigator — NIMS
Locations (1):
- Dr. Raghunathrao, Hyd, Andhra Pradesh, India